CLINICAL TRIAL: NCT01393015
Title: Using a Closed-loop System for Oxygen Delivery (FreeO2) to Optimize Oxygentherapy in Patients With Exacerbations of Chronic Obstructive Pulmonary Disease.
Brief Title: Using a Closed-loop System for Oxygen Delivery (FreeO2) to Optimize Oxygentherapy in Patients With COPD Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: François Lellouche, MD, CRIUCPQ
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FreeO2-COPD-5ePC
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-05

CONDITIONS: COPD Exacerbation
Keywords: automatic; automation; oxygen; weaning; COPD; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FreeO2 system (Experimental): FreeO2 is a new system that automatically adjusts the oxygen flow delivered to patients in closed-loop based on the SpO2 signal. This system is intended to maintain SpO2 in a predefined target and to adapt oxygen flow to patient's needs.
  Interventions: Device: Automated settings on the oxygen delivery device
- Rotameter (flowmeter) (Active Comparator): A rotameter is a device that measures the flow rate of liquid or gas in a closed tube.
  Interventions: Device: Manual settings with FreeO2 system in collection mode

INTERVENTIONS:
Device: Automated settings on the oxygen delivery device — FreeO2 automatically adjusts the oxygen flow delivered to patients based on the SpO2 signal. Patients keep using the same device for duration of hospitalization.
  Arms: FreeO2 system
Device: Manual settings with FreeO2 system in collection mode — Oxygen flow delivery is adjust by nurse and respiratory therapists. Standard medical treatment. Patients keep using the same device for duration of hospitalization.
  Arms: Rotameter (flowmeter)

SUMMARY:
Aim: The purpose of this study is to evaluate the use feasibility of FreeO2 so as to deliver automatically oxygen and to enable a remote medical monitoring with a homogeneous patient population hospitalize for Chronic obstructive pulmonary disease (COPD)exacerbation.

Hypothesis: The principal hypothesis is that FreeO2 is possible and well-accepted by nurses and medical personnel and there are advantages to use this system. In comparison with the common oxygen delivery (the rotameter), the hypothesis is that FreeO2 system will make for a better control of the oxygen saturation in function of designed target, reducing the desaturation time and hyperoxia. We think that oxygen weaning will be faster than classical way if it is automated. In addition, FreeO2 could reduce the number of intervention by nurse personnel and to improve the support with centralized monitoring in the FreeO2 group.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for COPD exacerbation
* 40 Years and older
* Former or current smoker greater than or equal to 10 pack-years
* Suspicion or diagnosis of COPD at the hospitalisation
* Acute dyspnea or acute aggravation of dyspnea
* Respiratory rate greater than or equal to 20 breaths/min
* Patient needs an oxygen therapy by nasal cannula with oxygen delivered between 0.5 to 8L/min to hold SpO2 greater than or equal to 92%

Exclusion Criteria:

* Imminent indications for intubation
* FreeO2 system is unavailable at the moment of randomization
* Patient in isolation (barrier nursing) to the inclusion
* Patient participates to another clinical trial without possibility of co-enrollment
* Patient with diagnosis of sleep apnea

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Possibility to use a new closed-loop system for oxygen delivery in common practice | 6 months
  We will see if nurses and medical personnel are agree to work with FreeO2 system. We want to know if the new system of automated adjustment of oxygen flow is useful in common practice.

SECONDARY OUTCOMES:
Time of oxygen weaning between common oxygen delivery and closed-loop automatic titration of oxygen flow based on SpO2. | 6 months
Percentage of time with desaturation during the oxygentherapy | 6 months
Percentage of time with hyperoxia during the oxygentherapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, Md, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Centre de recherche de l'institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Poder TG, Kouakou CRC, Bouchard PA, Tremblay V, Blais S, Maltais F, Lellouche F. Cost-effectiveness of FreeO2 in patients with chronic obstructive pulmonary disease hospitalised for acute exacerbations: analysis of a pilot study in Quebec. BMJ Open. 2018 Jan 23;8(1):e018835. doi: 10.1136/bmjopen-2017-018835. PMID 29362258